CLINICAL TRIAL: NCT05171725
Title: Multidisciplinary Expert System for the Assessment & Management of Complex Brain Disorders
Acronym: MES-CoBraD
Status: Recruiting | Type: Observational
Sponsor: Neurological Institute of Athens (Other)
Collaborators: Rabin Medical Center (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); King's College London (Other); Uppsala University (Other); Holistic IKE (Unknown); National Technical University of Athens (Other); Evolution Projects (Unknown); Engineering Ingegneria Informatica S.p.A. (Unknown); SOFTWARE IMAGINATION & VISION SRL (Unknown); Vrije Universiteit Brussel (Other); STICHTING LIBER (Unknown); University of Edinburgh (Other); CyberEthics Lab. srls (Unknown)
Responsible Party: Sponsor
Other Study IDs: EU-Horizon-2020-965422
Record Dates: First submitted 2021-09-30; First posted 2021-12-29 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Dementia; Alzheimer Disease; Epilepsy; Sleep Disorder; Circadian Rhythm Disorders; Healthy
Keywords: artificial intelligence; expert systems; deep-phenotyping
MeSH Terms: conditions — Dementia; Alzheimer Disease; Epilepsy; Sleep Wake Disorders; Chronobiology Disorders | interventions — Blood Specimen Collection; Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood (plasma and serum) and CSF biosamples collected and retained in deep freeze.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sleep and Circadian Disorders: Observational deep phenotyping of people presenting with Sleep and Circadian disorders. Participants will undergo a comprehensive multidisciplinary protocol of clinical assessment by an expert clinician, neuropsychological testing by a neuropsychologist through paper-and-pencil and tablet tests, actigraphy, polysomnography with concurrent electroencephalography, pre- and post- sleep cognitive testing and biosample acquisition, and where available provide access to wearable data, therapeutic device data (e.g., PAP/NIV), and brain imaging
  Interventions: Diagnostic Test: EEG,PSG; Diagnostic Test: biosample collection (blood and CSF); Diagnostic Test: neuropsychological testing; Diagnostic Test: actigraphy; Diagnostic Test: clinician assessment
- Neurocognitive Disorders: Observational deep phenotyping of people presenting with Dementia (including Alzheimer's disease, vascular disease, frontotemporal dementia). Participants will undergo a comprehensive multidisciplinary protocol of clinical assessment by an expert clinician, neuropsychological testing by a neuropsychologist through paper-and-pencil and tablet tests, actigraphy, polysomnography with concurrent electroencephalography, pre- and post- sleep cognitive testing and biosample acquisition, and where available provide access to wearable data, therapeutic device data (e.g., PAP/NIV), and brain imaging
  Interventions: Diagnostic Test: EEG,PSG; Diagnostic Test: biosample collection (blood and CSF); Diagnostic Test: neuropsychological testing; Diagnostic Test: actigraphy; Diagnostic Test: clinician assessment
- Epilepsy disorders: Observational deep phenotyping of people presenting with seizures and Epilepsy disorder. Participants will undergo a comprehensive multidisciplinary protocol of clinical assessment by an expert clinician, neuropsychological testing by a neuropsychologist through paper-and-pencil and tablet tests, actigraphy, polysomnography with concurrent electroencephalography, pre- and post- sleep cognitive testing and biosample acquisition, and where available provide access to wearable data, therapeutic device data (e.g., PAP/NIV), and brain imaging
  Interventions: Diagnostic Test: EEG,PSG; Diagnostic Test: biosample collection (blood and CSF); Diagnostic Test: neuropsychological testing; Diagnostic Test: actigraphy; Diagnostic Test: clinician assessment
- Healthy controls: Participants will undergo a comprehensive multidisciplinary protocol of clinical assessment by an expert clinician, neuropsychological testing by a neuropsychologist through paper-and-pencil and tablet tests, actigraphy, polysomnography with concurrent electroencephalography, pre- and post- sleep cognitive testing and biosample acquisition, and where available provide access to wearable data, therapeutic device data (e.g., PAP/NIV), and brain imaging
  Interventions: Diagnostic Test: EEG,PSG; Diagnostic Test: biosample collection (blood and CSF); Diagnostic Test: neuropsychological testing; Diagnostic Test: actigraphy; Diagnostic Test: clinician assessment

INTERVENTIONS:
Diagnostic Test: EEG,PSG — concurrent overnight sleep study with full electroencephalography (in-lab or at home)
Diagnostic Test: biosample collection (blood and CSF) — blood or CSF collection for analyses of neurodegenerative, inflammatory, and, per condition, genetic information
Diagnostic Test: neuropsychological testing — paper and pencil, as well as tablet based cognitive testing
Diagnostic Test: actigraphy — week long actigraphy assessment with concurrent sleep diary acquisition
Diagnostic Test: clinician assessment — standard clinical assessment by an expert clinician in the respective field of brain disorders

SUMMARY:
The Multidisciplinary Expert System for the Assessment & Management of Complex Brain Disorders (MES-CoBraD) is an interdisciplinary project combining Real-World Data (RWD) from multiple clinical and consumer sources through comprehensive, cost-efficient, and fast protocols towards improving diagnostic accuracy and therapeutic outcomes in people with Complex Brain Disorders (CoBraD), as reflected in Neurocognitive (Dementia), Sleep, and Seizure (Epilepsy) disorders and their interdependence. It brings together internationally recognized experts in medicine, engineering, computer science, social health science, law, and marketing and communication from across Europe, and combines clinical information and scientific research in CoBraD with technical innovation in secure data-sharing platforms, artificial intelligence algorithms, and expert systems of precision and personalized care, with a primary focus on improving the quality of life of patients, their caregivers, and the society at large. It leverages RWD from diverse CoBraD populations across cultural, socioeconomic, educational, and health system backgrounds, with special attention on including vulnerable populations and minorities in an equitable manner and engaging key stakeholders to maximize project impact.

ELIGIBILITY:
Inclusion Criteria:

* All participants willing to undergo comprehensive assessment who visit one of three clinics (Epilepsy, Neurocognitive disorders, and Sleep Disorders), and healthy volunteers

Exclusion Criteria:

* participant disinterest

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study aims to develop an Expert System for the assessment and management of complex brain disorders in real-world practice and participants who present in all of the above clinics are eligible, in order to obtain data as close to real-world practice as possible.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Expert System Accuracy for the Assessment of Complex Brain Disorders | 3 years
  Pursuing external cross-validation using training and test sample data acquired during MES-CoBraD, examine the sensitivity, specificity, accuracy, and likelihood ratios in making an accurate diagnosis of Complex Brain Disorders (neurocognitive, epilepsy, sleep disorders), compared to gold standard diagnostic criteria.
Expert System Accuracy for the Management of Complex Brain Disorders | 3 years
  Pursuing external cross-validation using training and test sample data acquired during MES-CoBraD, examine the sensitivity, specificity, accuracy, and likelihood ratios in recommending standard of care treatment decisions in Complex Brain Disorders (neurocognitive, epilepsy, sleep disorders), compared to gold standard professional society recommendations.

SECONDARY OUTCOMES:
Examine safety of approved therapies for Complex Brain Disorders | 3 years
  Test for statistically significant Side-Effect differences within 6 months of initiating approved treatments for Complex Brain Disorders between participants receiving and not receiving disease-specific therapies. Side effect reporting will be combined from patient, caregiver, and clinician input. Side effects are defined by a combination of predefined common and significant side-effect options and free text.
Prevalence co-occurrence of Complex Brain Disorders (Neurocognitive, Sleep, and Epilepsy disorders) | 3 years
  Within each of the three types of CoBraD, examine the frequency of comorbidity of the other two following comprehensive diagnostic protocols
Examine efficacy of approved therapies for Complex Brain Disorders | 3 years
  Test for statistically significant efficacy differences of using approved treatments for Complex Brain Disorders over the 3 year period of the study, between participants receiving and not receiving disease-specific therapies post sample stratification. Efficacy data will be combined from patient, caregiver, and clinician input according to the respective CoBraD efficacy outcome measures (e.g., MoCA for neurocognitive, seizure frequency and severity for epilepsy, PSQI for sleep disorders).

CONTACTS AND LOCATIONS:
Overall Officials: Elissaios Karageorgiou, Study Director — Neurological Institute of Athens; Ioannis Stavropoulos, Study Director — King's College London; Ophir Keret, Study Director — Rabin Medical Center; Juan Fortea, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (4):
- Neurological Institute of Athens, Athens, Greece
- Rabin Medical Center, Petah Tikva, Israel
- Sant Pau Memory Clinic, Barcelona, Spain
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and depersonalized on a local site repository, and then uploaded in the secure MES-CoBraD Platform. An estimated six months after study completion, data will be made available to other researchers through the MES-CoBraD Platform.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: an estimated 6 months after study completion
Access Criteria: These will be developed upon completion of the Platform. The platform will contain both opensource and pre-existing proprietary code, and some of the code will not be made available to researchers, but will be functional on the Platform.

REFERENCES:
- See also: Study site — http://mes-cobrad.eu